CLINICAL TRIAL: NCT04056403
Title: The Use of Ultrasound to Evaluate Precision and Analgesic Efficacy of Labor Epidural Analgesia
Brief Title: Ultrasound Evaluation of Labor Epidural
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201907006RINC
Record Dates: First submitted 2019-08-07; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Parturient
Keywords: labor epidural; ultrasound

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To compare the labor epidural analgesic (EA) profiles between landmark insertion EA levels which are congruent and ingruent to ultrasound confirmation in lateral decubitus position.

DETAILED DESCRIPTION:
Epidural analgesia is the mainstream method for labor analgesia. Landmark identification of L3 to L5 spinous process is most commonly applied for determination of epidural insertion. However, the precision of epidural catheter insertion site was affected by physiological and anatomical variations in pregnant women and positions such as sitting or lateral decubitus. Previous study showed the clinical estimation would be ≥ 1 vertebral level higher than the anatomical position determined by ultrasound at least 40% of the time in sitting position among western pregnant women. For asian parturients, epidural analgesia is commonly performed in lateral decubitus position because of smaller stature. In addition, it remains uncertain whether the landmark epidural insertion level congruent or ingruent is associated with different analgesia profiles such as the dosage requirement and the frequncy of adjustment.

ELIGIBILITY:
Inclusion:

1. Normal spontaneous delivery parturients receiving labor epidural analgesia in first stage of labor
2. Using patient-controlled epidural analgesia

Exclusion:

1. who has an accidental epidural puncture
2. who receives epidural insertion by ultrasound identification
3. who uses of magnesium sulfate

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Parturient who receive labor epidural
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Accuracy of landmark epidural level | 10 minute
  Validation of landmark localization of epidural insertion level by using ultrasound examination

SECONDARY OUTCOMES:
Labor analgesic dose | one day
  Influences of accurate epidural insertion level on labor epidural analgesic dose

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan